CLINICAL TRIAL: NCT03057938
Title: Subjects With Subjective Cognitive Decline: 18F-Florbetaben Positron Emission Tomography Study
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The sponsor cannot provide the study treatment
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Principal Investigator, Anna Cruceta, Project Manager, Fundacion Clinic per a la Recerca Biomédica
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Euro-SCD-FBB2
Record Dates: First submitted 2017-02-15; First posted 2017-02-20 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2024-03

CONDITIONS: Subjective Cognitive Decline
Keywords: Alzheimer; Subjective Cognitive Decline; Florbetaben
MeSH Terms: interventions — 4-(N-methylamino)-4'-(2-(2-(2-fluoroethoxy)ethoxy)ethoxy)stilbene

STUDY DESIGN:
Intervention Model Description: Phase II, open-label clinical trial with a medicinal product.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 18F-Florbetaben (FBB) (Experimental): 18F-Florbetaben
  Interventions: Drug: 18F-Florbetaben (FBB)

INTERVENTIONS:
Drug: 18F-Florbetaben (FBB) — All participants will receive a single intravenous dose of 300 MBq of FBB followed by PET scan.
  Other Names: FBB

SUMMARY:
Phase II, open-label clinical trial with a medicinal product. A total of 30 subjects will be included in the study.

All participants will receive a single intravenous dose of 300 MBq of FBB. A 20-minute PET image should be acquired starting at approximately 90 minutes after intravenous injection of FBB.

The present proposal aims are: to assess safety of a single dose of FBB followed by PET scan in individuals with subjective cognitive decline (SCD), to determine the number of SCD subjects with positive visual FBB-PET scan, to determine the number of SCD subjects with positive standardized uptake value ratios (SUVRs) of FBB-PET scan and to explore the cortical pattern of amyloid deposition in SCD subjects.

DETAILED DESCRIPTION:
statistical methods: Primary outcomes For the analysis of the primary outcomes, a descriptive statistical approach will be implemented, calculating the proportion of adverse events and the proportion of SCD subjects that are positive for FBB-PET at visual assessment 9.2 Data Management Demographical and neuropsychological data will be entered in a data base. Statistical analyses will be performed with the SPSS software for Windows (v.22.0).

Sample size A sample size of 30 subjects has been estimated. Since this is a proof-of-concept study, this assumption has been based on previously published data.

Statistical significance and adjustments for multiplicity The analysis will be carried out according to the principles of the ICHE9 Guide and in accordance with the recommendations of CPM/EWP/908/99 Points to Consider on Multiplicity issues in Clinical Trials. The contrast will be carried out with an Error of Type 5 bilateral I. In any case, since this is a exploratory study, there will be no adjustments for multiplicity.

Criteria for discontinuation

The study will be completed when these two premises are met:

* Inclusion of the number of patients needed for the sample size
* End of clinical monitoring No interim analyses are planned.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be committed to participate and complete all study procedures.
* The patient must report a memory problem (in isolation or in combination with complaints in other domains) with concern.
* Age ≥ 60
* Mini-Mental State Examination cutoff for inclusion will be ≥ 26.
* Clinical Dementia Rating <0,5.
* Subjects must have signed the Informed Consent Form voluntarily to participate in the study.

Exclusion Criteria:

* Subjects those are not able to complete the study.
* Any major disease or history of a major disease, especially hepatobilliar disease (AST /ALT ≥ 5 x ULN) or advanced renal insufficiency (creatinine ≥ 2 x ULN).
* Current or previous history of alcohol abuse or epilepsy.
* Allergic to Florbetaben or any of its constituents.
* Multiple drug allergies and/or previous history of contrast allergy.
* Any disease or history of disease which, in the opinion of the investigator, can cause disturbance of brain function (e.g. vitamin B12 or folic acid deficiency, disturbed thyroid function).
* Evidence for any other neurological or psychiatric disease, eg. parkinsonism, history of stroke or seizure.
* Pregnancy or breast feeding or planned pregnancy during the study period.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | 24 months
  Incidence of Adverse events of a single dose of FBB followed by PET scan in individuals with Subjective Cognitive Decline
Positive visual FBB-PET scan | 24 months
  Proportion of Subjective Cognitive Decline subjects that present positive uptake after FBB-PET through visual examination.

SECONDARY OUTCOMES:
Positive standardized uptake value ratios | 24 months
  Proportion of SCD subjects presenting standardized uptake value ratios (SUVRs) of FBB-PET higher than 1,4.
Cortical pattern of amyloid deposition | 24 months
  To explore the cortical pattern of amyloid deposition in SCD subjects at visual and semi-quantitative examination.

CONTACTS AND LOCATIONS:
Overall Officials: Lorena Rami, Dr, Principal Investigator — Fundació Clinic